CLINICAL TRIAL: NCT02629380
Title: Early Viscosupplementation After Partial Meniscectomy: a Double Blind, Placebo Controlled Randomized Trial
Brief Title: Early Viscosupplementation After Partial Meniscectomy: a Randomized Controlled Trial
Acronym: HA-MEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Federica Balboni, BScD, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rizzoli HA-MEN
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Meniscus Lesion
Keywords: meniscectomy; hyaluronic acid; intra-op injection; randomized controlled trial; placebo
MeSH Terms: interventions — Hyaluronic Acid; Meniscectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyaluronic acid group (Experimental): Single injection of 3 ml HA (Hymovis, Fidia Farmaceutici SpA, Padova, Italy) at the end of the arthroscopic meniscectomy
  Interventions: Biological: hyaluronic acid
- meniscectomy alone (Other): Arthroscopic meniscectomy alone
  Interventions: Procedure: meniscectomy alone

INTERVENTIONS:
Biological: hyaluronic acid — A single injection of 3 ml hyaluronic acid to be performed under arthroscopic view at the end of meniscectomy
  Arms: Hyaluronic acid group
Procedure: meniscectomy alone — The patients randomized in this group will receive arthroscopic meniscectomy alone
  Arms: meniscectomy alone

SUMMARY:
The rational of intra-articular viscosupplementation is based on both the biological and mechanical properties of HA, which exerts positive effects on the modulation of the entire joint environment.

The aim of the present double blind controlled study was to evaluate the effects in terms of pain control and functional recovery provided by a single intra-operative injection of HA performed at the end of arthroscopic partial meniscectomy.

Patients included in this trial were randomized in two treatment groups: the first one received a single injection of HA (Hymovis 24 mg/3ml, Fidia Farmaceutici Spa, Padova, Italy) at the end of the arthroscopic meniscectomy, whereas the second group was treated by surgery alone.

All patients were evaluated basally, at 15, 30, 60, and 180 days after surgery by the following evaluation tools: IKDC (International Knee Documentation Committee) subjective, VAS (Visual Analogue Score) for pain, EQ-VAS for general Health Status, KOOS (Knee Injury and Osteoarthritis Outcome Score) and Tegner score. Furthermore, during the basal evaluation and at each follow-up visit up to 2 months, active and passive Range of Motion (ROM) of both the operated and contralateral knee were documented; also in addition, the trans-patellar circumference of both knees was registered to assess the trend of knee swelling over time.

ELIGIBILITY:
Inclusion Criteria:

1. chronic symptomatic meniscal tears requiring partial resection;
2. healthy contra-lateral knee (i.e. no pain or functional limitation in the contra-lateral joint);

Exclusion Criteria:

1. previous surgery on the index knee;
2. other concurrent articular lesion requiring surgical treatment (e.g.: cartilage or ligament injuries);
3. history of knee infectious arthritis;
4. concurrent rheumatic, metabolic or severe systemic disease;
5. Body Mass Index (BMI) > 30;
6. known hypersensibility or allergy to/towards HA ;
7. alcohol or other substances abuse/excess.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in IKDC (International Knee Documentation Committee) score | basal, 15,30,60,180 days

SECONDARY OUTCOMES:
Change in KOOS (Knee Injury and Osteoarthritis Outcome Score) | basal, 15,30,60,180 days
Change in Tegner Score | basal, 15,30,60,180 days
Change in VAS (Visual Analogue Scale) for pain | basal, 15,30,60,180 days
Change in EQ-VAS for general health | basal, 15,30,60,180 days
Change in transpatellar circumference over time | basal, 15,30,60,180 days
Change in active and passive ROM | basal, 15,30,60,180 days
Adverse events report | 15 days
Adverse events report | 30 days
Adverse events report | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator — II Clinic and Nano-biotechnology Lab, Rizzoli Orthopedic Institute, Bologna, Italy
Locations (1):
- II Orthopaedic Clinic, Rizzoli Orthopaedic Institute, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edouard P, Rannou F, Coudeyre E. Animal evidence for hyaluronic acid efficacy in knee trauma injuries. Review of animal-model studies. Phys Ther Sport. 2013 May;14(2):116-23. doi: 10.1016/j.ptsp.2013.02.001. Epub 2013 Mar 16. PMID 23506791
- [Background] Freymann U, Endres M, Goldmann U, Sittinger M, Kaps C. Toward scaffold-based meniscus repair: effect of human serum, hyaluronic acid and TGF-ss3 on cell recruitment and re-differentiation. Osteoarthritis Cartilage. 2013 May;21(5):773-81. doi: 10.1016/j.joca.2013.02.655. Epub 2013 Mar 5. PMID 23473977
- [Background] Thein R, Haviv B, Kidron A, Bronak S. Intra-articular injection of hyaluronic acid following arthroscopic partial meniscectomy of the knee. Orthopedics. 2010 Oct 11;33(10):724. doi: 10.3928/01477447-20100826-11. PMID 20954664
- [Background] Tan GK, Dinnes DL, Butler LN, Cooper-White JJ. Interactions between meniscal cells and a self assembled biomimetic surface composed of hyaluronic acid, chitosan and meniscal extracellular matrix molecules. Biomaterials. 2010 Aug;31(23):6104-18. doi: 10.1016/j.biomaterials.2010.04.018. Epub 2010 May 14. PMID 20471080
- [Background] Westrich G, Schaefer S, Walcott-Sapp S, Lyman S. Randomized prospective evaluation of adjuvant hyaluronic acid therapy administered after knee arthroscopy. Am J Orthop (Belle Mead NJ). 2009 Dec;38(12):612-6. PMID 20145786
- [Background] Waddell DD, Bert JM. The use of hyaluronan after arthroscopic surgery of the knee. Arthroscopy. 2010 Jan;26(1):105-11. doi: 10.1016/j.arthro.2009.05.009. Epub 2009 Nov 25. PMID 20117634
- [Background] Cake M, Read R, Edwards S, Smith MM, Burkhardt D, Little C, Ghosh P. Changes in gait after bilateral meniscectomy in sheep: effect of two hyaluronan preparations. J Orthop Sci. 2008 Nov;13(6):514-23. doi: 10.1007/s00776-008-1279-6. Epub 2008 Dec 17. PMID 19089539
- [Background] Mathies B. Effects of Viscoseal, a synovial fluid substitute, on recovery after arthroscopic partial meniscectomy and joint lavage. Knee Surg Sports Traumatol Arthrosc. 2006 Jan;14(1):32-9. doi: 10.1007/s00167-005-0625-x. Epub 2005 May 26. PMID 15918064
- [Derived] Filardo G, Di Matteo B, Tentoni F, Cavicchioli A, Di Martino A, Lo Presti M, Iacono F, Kon E, Marcacci M. No Effects of Early Viscosupplementation After Arthroscopic Partial Meniscectomy: A Randomized Controlled Trial. Am J Sports Med. 2016 Dec;44(12):3119-3125. doi: 10.1177/0363546516660070. Epub 2016 Aug 15. PMID 27528611